CLINICAL TRIAL: NCT03765697
Title: An Open-label, Multicenter, Multiple-dose, Phase III Study With Lidocaine 5% Medicated Plaster in Patients Suffering From Postherpetic Neuralgia
Brief Title: A Study With Lidocaine 5% Medicated Plaster in Patients Suffering From Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF10004/02
Record Dates: First submitted 2018-11-27; First posted 2018-12-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Post Herpetic Neuralgia
Keywords: post-herpetic neuralgia; lidocaine
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Lidocaine; Lidoderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lidocaine 5% medicated plaster (Experimental): Up to 3 plasters were applied per day.
  Interventions: Drug: Lidocaine 5% medicated plaster

INTERVENTIONS:
Drug: Lidocaine 5% medicated plaster — Topical application at the site of skin affected by painful PHN for up to 12 hours per day (plaster-free interval at least 12 hours).
  Other Names: Versatis (Trade Mark); Neurodol Tissugel (Trade Mark); Lidoderm (Trade Mark)

SUMMARY:
This study was performed to evaluate the local and systemic safety profile and the analgesic efficacy of long-term treatment with lidocaine 5% medicated plaster (Lido-Patch).

The study was an open-label, multi-center, multiple-dose, Phase III study and comprised a main and an extension period. 161 participants who completed treatment in KF10004/01 (NCT03745404) and 98 newly recruited participants were enrolled.

DETAILED DESCRIPTION:
The main period was performed in 34 sites in 12 European countries (259 participants). Treatment duration was up to 12 months. All participants applied lidocaine 5% medicated plaster (containing 700 mg lidocaine per plaster) topically at the site of the skin affected by painful PHN. Depending on the size of the affected skin area, up-to 3 plasters were simultaneously applied for up to 12 hours per day (with a plaster-free interval of at least 12 hours). Study objectives of the main period were to evaluate the local and systemic safety profile and the analgesic efficacy of lidocaine 5% medicated plaster, and to evaluate the pharmacokinetics of lidocaine and its metabolite 2,6-xylidine in the target population after multiple administrations of lidocaine 5% medicated plaster by means of population kinetics. The study results were planned to be evaluated descriptively.

102 participants who were satisfied with the treatment in the main study period entered the open-label extension period with continued treatment. 27 sites in 12 countries participated in the extension period. Enrollment in the extension period coincided with last visit of the main period of the study. Treatment duration was up to 4.4 years in the extension period. The objective of the extension period was to evaluate the long-term local and systemic safety profile and the long-term analgesic efficacy of treatment with lidocaine 5% medicated plaster in the subpopulation who had completed 12 months of treatment in the open-label main study period.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, male and female, with a minimum age of 50 years at screening.
* Participants who had postherpetic neuralgia (PHN) for at least 3 months after healing of a herpes zoster skin rash.
* Only for patients who had not participated in the KF10004/01 (NCT03745404) study: Pain score of at least 4, based on an 11-point numerical rating scale (NRS) (scale of 0-10), at the screening visit. The pain assessment is the participant's recall of the pain intensity since the previous week.
* Written informed consent given.

Exclusion Criteria:

* Participation in another study of investigational drugs or devices parallel to, or less than 30 days before screening, or previous participation in this study, except previous participation in the KF10004/01 study.
* Known to or suspected of not being able to comply with the study protocol.
* Any clinically significant condition that would, in the investigator's opinion, preclude study participation for instance alcohol, medication or drug dependency, neurotic personality, psychiatric illness, epilepsy or suicide risk.
* Pregnancy or nursing mother.
* Woman in childbearing age without satisfactory contraception.
* Hypersensitivity to lidocaine or amide-type local anesthetic drugs.
* Active herpes zoster lesion or dermatitis of any origin at the affected site with PHN.
* Evidence of another cause for pain in the area affected by herpes zoster in addition to PHN, such as lumbar radiculopathy, surgery or trauma, if this could confound assessment or self-evaluation of the pain due to PHN.
* Participants who had neurological ablation by block or neurosurgical intervention for control of pain in PHN.
* Participants using topically applied analgesic compounds on the PHN affected area.
* Presence of other severe pain that could confound assessment or self-evaluation of the pain due to PHN.
* Participants with severe hepatic disorder and/or alanine or aspartate aminotransferase equal to or above 3-fold the upper limit of normal (ULN).
* Participants with severe renal disorder and/or increased serum creatinine equal to or above 1.5-fold the upper limit of normal (ULN).
* Participants who are undergoing active treatment for cancer, are known to be infected with the human immunodeficiency virus (HIV), or being acutely and intensively immunosuppressed following transplantation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2003-07-16 (Actual); Primary Completion 2005-07-12 (Actual); Study Completion 2009-02-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (main study period) | From first plaster application up to 12 months
  Treatment emergent adverse events (TEAEs) were continually monitored through the main period of the study (12 months). Incidences were calculated based on all events reported up to 12 months. No primary endpoint was defined for this study.

SECONDARY OUTCOMES:
Pain relief (main study period): verbal rating scale | After 1, 6, 12, 18, 26, 34, 42, and 52 weeks (or early withdrawal)
  Pain relief was assessed starting 1 week (new participants) or 6 weeks after treatment initiation (participants from KF10004/01) until the final visit of the main study period. The average pain relief during the last week before the visit was assessed using a 6-item verbal rating scale (VRS) with categories 1 = worse, 2 = no pain relief, 3 = slight, 4 = moderate, 5 = a lot, and 6 = complete.
Pain intensity (main study period): Numeric Rating Scale | At screening/enrollment and after 1, 6, 12, 18, 26, 34, 42, and 52 weeks (or early withdrawal)
  The participant's recall of worst, least, and average pain intensity in the last week prior to each visit were assessed using an 11-point Numeric Rating Scale (NRS from 0 = no pain to 10 = pain as bad as you can imagine).
Pain relief (extension period): verbal rating scale | Every 6 months after first plaster application in the extension period up to 4.4 years (or early withdrawal)
  The participant's recall of average pain relief during plaster application in the last week prior to each visit in the extension period was assessed using a 6-item VRS with categories 1 = worse, 2 = no pain relief, 3 = slight, 4 = moderate, 5 = a lot, and 6 = complete.
Number of participants with treatment emergent adverse events (extension period) | Every 6 months after first plaster application in the extension period up to 4.4 years (including a follow-up visit 1-2 weeks after last regular 6-month visit or early withdrawal)
  Treatment emergent adverse events were continually monitored for or asked about at each visit scheduled every 6 months in the extension period. The extension period lasted for up to 4.4 years and included a follow-up visit (1-2 weeks after last regular 6-month visit [or early withdrawal]). Adverse event incidences were calculated based on all events reported in the extension period.

OTHER OUTCOMES:
Allodynia severity rating (main study period) | At screening/enrollment, and after 1, 6, 12, 18, 26, 34, 42, and 52 weeks (or early withdrawal)
  Allodynia severity was rated using the following categorical scale: 0 = no pain or discomfort to touch; 1 = uncomfortable, but tolerable to touch; 2 = painful; 3 = extremely painful, participant cannot stand touching. The test was conducted by means of a brush (type N12). The painful PHN area was stroked with the brush and the intensity of allodynic pain was assessed by the participant.
Clinical Global Impression of Change (CGIC) (main study period) | At 26 weeks of treatment in the main study period and at the final visit (at 52 weeks, or early withdrawal)
  Investigators were asked to describe their overall impression of the change of the participant's condition/pain by answering the following question: "Compared to the patient's condition at admission to the project, how much has he/she changed?" The categorical scale comprises the categories not assessed = 0, very much improved = 1, much improved = 2, minimally improved = 3, no change = 4, minimally worse = 5, much worse = 6, and very much worse = 7.
Short Form-36 Quality of Life Index (SF-36) (main study period) | At screening, and after 12, 26, 42, and 52 weeks (or early withdrawal)
  The Short Form 36 Quality of Life Index (SF-36 [Trade Mark]) standard version with a 4-week recall period was used as a self-assessment.
  Eleven questions were answered on binomial (Yes/No) or on 3-, 5-, or 6-point categorical scales to generate the 8 raw scales (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health). Higher values of the raw scales represent a better outcome. The raw scales were converted into a transformed scale (transformed scale = [(actual raw score - lowest possible raw score) / possible raw score range] x 100).
Short Form McGill Pain Questionnaire (SF-MPQ) (main study period) | At screening, and after 12, 26, 42, and 52 weeks (or early withdrawal)
  The SF-MPQ includes 15 words (11 sensory, 4 affective). Each word or phrase is rated on a 4-point intensity scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe). In addition, the 6-point Present Pain Intensity (PPI) rating (no pain, mild, discomforting, distressing, horrible, excruciating) is included as is a visual analogue scale for rating pain intensity. Total score as well as sensory and affective sub-scores were calculated.
Clinical Global Impression of Change (CGIC) (extension period) | Every 6 months after first plaster application in the extension period up to 4.4 years (or early withdrawal)
  Investigators were asked to describe their overall impression of the change of the participant's condition/pain by answering the following question: "Compared to the patient's condition at admission to the project, how much has he/she changed?" (categories: not assessed = 0, very much improved = 1, much improved = 2, minimally improved = 3, no change = 4, minimally worse = 5, much worse = 6, very much worse = 7).
Patient's Global Impression of Change (PGIC) (extension period) | Every 6 months after first plaster application in the extension period up to 4.4 years (or early withdrawal)
  Participants were asked to describe their overall impression of change of their condition/pain by answering the following question: "Compared to your pain at admission to the project, how much has it changed?" (categories: not assessed = 0, very much improved = 1, much improved = 2, minimally improved = 3, no change = 4, minimally worse = 5, much worse = 6, very much worse = 7).
Investigator's Global Evaluation of the IMP (extension period) | Every 6 months after first plaster application in the extension period up to 4.4 years (or early withdrawal)
  The assessment of the investigational medicinal product (IMP) was made on a 5-point categorical scale (poor, fair, good, very good, excellent). Investigators responded to the following question: "How would you rate the study medication the patient received for pain?"
Patient's Global Evaluation of the IMP (extension period) | Every 6 months after first plaster application in the extension period up to 4.4 years (or early withdrawal)
  The assessment of the IMP was made on a 5-point categorical scale (poor, fair, good, very good, excellent). Participants responded to the following question: "How would you rate the study medication you received for pain?"
Change in concomitant medication (main and extension period) | At enrollment into main study period; at last assessment in extension period (up to 5.4 years after enrollment)
  For each participant, the number of different medications taken for PHN symptoms was determined at enrollment into the and at the last assessment in the study. Participants were classified into 5 groups: 0, 1, 2, 3, and more than 3 different substances taken. Shifts were determined for enrollment to last assessment in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hans G, Sabatowski R, Binder A, Boesl I, Rogers P, Baron R. Efficacy and tolerability of a 5% lidocaine medicated plaster for the topical treatment of post-herpetic neuralgia: results of a long-term study. Curr Med Res Opin. 2009 May;25(5):1295-305. doi: 10.1185/03007990902901368. PMID 19366301
- [Result] Sabatowski R, Hans G, Tacken I, Kapanadze S, Buchheister B, Baron R. Safety and efficacy outcomes of long-term treatment up to 4 years with 5% lidocaine medicated plaster in patients with post-herpetic neuralgia. Curr Med Res Opin. 2012 Aug;28(8):1337-46. doi: 10.1185/03007995.2012.707977. Epub 2012 Jul 18. PMID 22769236